CLINICAL TRIAL: NCT04450615
Title: Effects of a 5-week Core Training Program on Core Muscles' Imbalances
Brief Title: Core Exercises Effects on Muscle Imbalances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athanasios Ellinoudis (Other)
Responsible Party: Sponsor-Investigator, Athanasios Ellinoudis, Principal Investigator, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ERC-006/2020
Record Dates: First submitted 2020-06-25; First posted 2020-06-29 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Muscle Atrophy or Weakness; Muscle Contraction; Core Stability
MeSH Terms: conditions — Muscular Atrophy; Asthenia | interventions — Core Stability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (Experimental): The first part of the program aims in pelvic and hip mobility and includes the following exercises, glute bridge, single-leg glute bridge, side-lying clam, side plank and side plank with hip abduction, on stable surface.
  The second part consists of exercises for deep and superficial trunk muscles. In the first exercise the participants learn to activate the transversus abdominis muscle from the crook-lying position, by performing abdominal hollow. Other exercises include the front plank, trunk curl-up, trunk curl-up on stable surface and curl-up on unstable surface (Swiss ball).
  The third part of the program consists of exercises for strengthening the lumbar multifidus muscle. The participants will perform prone trunk extension, superman exercise, quadruped diagonal arm and leg lift, single leg supine bridge and supine bridge on unstable surface (Swiss ball).
  Interventions: Other: Core stability
- Control group (No Intervention): The participants of this group will follow their typical daily routine

INTERVENTIONS:
Other: Core stability — The exercise protocol consists of the following sets and repetitions, with a total duration of 5 weeks and a frequency of 3 sessions per week.
  Dynamic exercises: 2 sets of 10 to 15 repetitions (each side) Isometric exercises: 2 sets of 5 to 15 seconds (each side) Week 1- As mentioned above Week 2- Add 1 set Week 3 - Add 5 seconds and 5 repetitions Week 4 - Add 1 set Week 5- Add 5 seconds and 5 repetitions
  Arms: Training group

SUMMARY:
This study aims in investigating the effects of a core muscles' strengthening program on core muscles' atrophy and contraction ability. Twenty healthy adults recruited and randomly assigned to either a 5-week training group developed to activate and strengthen local trunk muscles or a control group. The training program includes isometric bridging exercises from various positions and dynamic exercises for lumbopelvic stability. Core muscles' thickness will be assessed at rest and contracting conditions, prior and after the intervention, using ultrasonography.

DETAILED DESCRIPTION:
A total of 136 male and female adults, members of local gyms, were initially invited for participation in the study after giving their written consent. After a second contact with the participants, forms regarding the inclusion and exclusion criteria were sent for completion.

Of the 136 that initially answered positively for participation, 62 did not meet the inclusion criteria, based on their reports and the clinical examination by a health professional. Of the remaining 74 participants, 32 were excluded because of previous low back pain incidents and other recent musculoskeletal injuries that led to rehabilitation, while 22 decided to not participate for personal reasons.

The remaining 20 participants were randomly allocated to either training group or intervention group, by a neutral, blinded investigator who had no involvement and was unaware of the study purposes. The intervention group will be trained and supervised by a certified fitness instructor in a gym class, who will be responsible for the correct execution of the exercises. The duration of the intervention will be 5 weeks, 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old
* Trained recreationally at least 2 times a week, for the past 3 years
* Healthy
* No musculoskeletal injuries in the 6 months prior to the study

Exclusion Criteria:

* History of chronic low back pain
* History of hip, pelvic or low back surgery
* History of acute low back pain with duration at least 1 week, the preceding 6 months
* Involvement in similar core stability training programs the last 12 moths prior to this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Transversus abdominis (TrA) muscle thickness at rest and contraction | Change from baseline assessment at 5 weeks
  Muscle thickness (mm) is measured using ultrasonography
Lumbar multifidus (LM) muscle thickness at rest and contraction | Change from baseline assessment at 5 weeks
  Muscle thickness (mm) is measured using ultrasonography

SECONDARY OUTCOMES:
Contraction thickness ratio (CTR) of TrA and LM muscle | Change from baseline assessment at 5 weeks
  This is calculated by subtracting rest thickness from contraction thickness, dividing it to rest thickness and multiplying this value by 100 [(contraction thickness-rest thickness/rest thickness)*100]

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Ellinoudis, PhD, Principal Investigator — Laboratory of Neuromechanics, Aristotle University of Thessaloniki
Locations (1):
- Laboratory of Neuromechanics, Department of physical education and sport sciences, Aristotle University of Thessaloniki, Serres, Greece

IPD SHARING:
Plan to Share IPD: No